CLINICAL TRIAL: NCT00956059
Title: Therapeutic Effect of Low-dose Prednisone Combined With MMF and FK506 in Focal Segmental Glomerulosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Gui Baosong, The Second Affiliated Hospital of Medical College,Xi'an JiaoTong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSX-090630-SAHXJTU; DBDZL-1; DX-FSGS-1; YW-JS-XX-TKMS; JL-5MG-50MG-500MG; JG-YX-1
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: focal segmental glomerulosclerosis; prednisone; mycophenolate mofetil; FK506
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Prednisone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prednisone, MMF and FK506 (Experimental)
  Interventions: Drug: prednisone, FK506, MMF
- prednisone (Active Comparator)
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone, FK506, MMF — 1.in the initial 3 months，prednisone dosage is 30mg per day；in the following 4~6 months，prednisone dose decreased to 20mg per day，then tapered gradually to 10mg per day；2.the initial dosage of FK506 is 0.2mg/kg/d, twice per day，the maintenance dosage is adjust to the serum concentration of FK506 (is maintained at the level of 6~10μg/L)；3. the initial dosage of MMF is 1.0g, twice per day，then reduce to 0.75 g, twice per day after 3 months
  Arms: prednisone, MMF and FK506
Drug: prednisone — In the initial 16~24 weeks，prednisone is given at full dose of 1mg/kg/d，then prednisone is tapered gradually，the whole course of treatment is 52 weeks
  Arms: prednisone

SUMMARY:
The aim of this clinical trial is to determine the effect and security of low-dose Prednisone Combined With MMF and FK506 in Focal Segmental Glomerulosclerosis.

DETAILED DESCRIPTION:
Focal segmental glomerular sclerosis (FSGS) is characterized by heavy proteinuria and nephritic syndrome in clinic. The major pathological change is scarring of the glomerulus that is focal and segmental. The incidence of FSGS is increasing in recent years, but no unified protocol for FSGS treatment has been provided. Corticosteroid is the primary drug for FSGS treatment in clinic. However, corticosteroid treatment has a low response rate as 20% in clinic but some severe side-effects. The side-effects of long-term corticosteroid treatment urged researchers to find more reliable and secure methods for FSGS treatment. The new immunosuppressants shed light on FSGS treatment recently. The usage of immunosuppressants to FSGS treatment is in the preliminary stage and accounts for a few problems. The main problems include the uncertainty of curative effects, the lack of large-scale clinical trial, the side-effects of long-term application, and the high recurrence rate after withdraw. FSGS is immune-induced damage, which includes abnormality of many steps in humoral immunity and cellular immunity. According to it, we designed to inhibit the immune response at multi-targets with Prednisone Combined With MMF and FK506. Thus the dosage of these drugs can be decreased to a secure level for long-term treatment while the side-effects can be controlled well. Prednisone Combined With MMF and FK506 then can be used to FSGS treatment with effectiveness and security.

ELIGIBILITY:
Inclusion Criteria:

* Urinary protein≥1.0g/24h
* Biopsy-proved FSGS
* Age≥16years
* Understanding of the content of this study，signing informed consent form
* Adherence to drug taking and being able to be long-term followed up

Exclusion Criteria:

* Sharp deterioration of renal function
* Refractory hypertension
* Secondary FSGS
* Serious disease of liver，active stage of viral hepatitis，or AST、ALT≥2.5 times of baseline
* Serious myelosuppression
* Being unable to be long-term followed up

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
proteinuria,serum protein,Scr,blood routine examination,liver function test,blood glucose and lipid test | 16~24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Baosong Gui, MD, Study Chair — The second affiliated hospital of Medical College, Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of medical college, Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732